CLINICAL TRIAL: NCT07397637
Title: KeySteps@JC Phase Two Parenting Program
Brief Title: A Strength-based Parenting Program for Parents With Young Children From 3 to 6 Years Old
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other); Education University of Hong Kong (Other); The Boys' and Girls' Clubs Association of Hong Kong (Other); Hong Kong Christian Service (Other); Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Anna Na Na Hui, Associate Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KeySteps@JCStrength-BasedStudy; 2022-0114-007 (Other Grant/Funding Number: Hong Kong Jockey Club Charities Trust)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Parenting Intervention
Keywords: Parenting, Strength-based, child-parent parallel design

STUDY DESIGN:
Intervention Model Description: The intervention study has four groups: a) the parenting program delivered in both school and hub, b) the parenting program delivered in school, c) the parenting program delivered in hub, and d) the parenting program to be delivered at a delayed timeframe.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parent-Child Parallel Program in school and hub (Experimental): It is an intervention for Parent-Child Parallel Program in both school and hub.
  Interventions: Behavioral: The Strength-based parenting program
- Parent-Child Parallel Program in school (Active Comparator): The program is delivered in school.
  Interventions: Behavioral: The Strength-based parenting program
- Parent-Child Parallel Program in hub (Active Comparator): The parenting program is delivered in hub.
  Interventions: Behavioral: The Strength-based parenting program
- Parent-Child Parallel Program with a delayed format (Active Comparator): The parenting program will be delivered in a delayed format
  Interventions: Behavioral: The Strength-based parenting program

INTERVENTIONS:
Behavioral: The Strength-based parenting program — A parenting program is designed with strength-based parenting theory and practice. It has 6 sessions for parents and young children when the children are at 3 years old, 4 sessions for them at 4 years old and another 4 sessions for them at 5 years old.

SUMMARY:
The parent education and family support component in phase 2 aims to strengthen protective factors of healthy child development and reduce risk factors of child abuse and neglect among disadvantaged families by providing community-based preventive interventions for children and their significant adults.

Participants include about 600 parents from randomly assigned 100 preschools to the four groups (group 1: hub + school support; group 2: school support; group 3: hub support; group 4: delay group).

The primary hypothesis is to examine the efficacy of the parenting programs for young children and their parents from K1 to K3. The programs are delivered by social workers at kindergartens or community hubs. The second aim/hypothesis of this project is to investigate the overall synergy impact of the community hub.

The success of the parent-child interactive program offers a foundation for the hub to further develop community-based parent education and family support programs that aim at building parents/caregivers' competence in optimizing child development and competence in caregivers and professionals through networking multiple ecological systems, i.e., family, school, and hub or other organizations in the community.

DETAILED DESCRIPTION:
Community hubs could be scaled up as a key setting where majority of intervention shall take place in to build capacity of significant others. For instance, there it will be an arena for the community-based parent education and family support programs. Community hubs act as a connector to bridge services. Due to disparity in resources and knowledge, parents in poverty may need extra rapport to bridge them to various supportive services available in the hub/community for the children's optimum development. This child and family centered approach can help foster community cohesion and raise family and children well-being.

The parenting program is designed with an emphasis on strength-based parenting practice and both children and parents have parallel sessions on the same character strength and also joint sessions to optimize the impact. Both quantitative and qualitative data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* parents whose children study in the 100 preschools taking part in the project

Exclusion Criteria:

* parents who do not give consent to take part

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in early parenting attitude | From enrollment to the end of treatment at 4-6 months
  1 indicates the lowest scores and 7 indicates the highest scores in affection and attachment between parents and children.
Change in strength-based parenting practice | From enrollment to the end of treatment at 6 months
  1 indicates lowest use of strength-based parenting practice and 7 indicates highest use of strength-based parenting practice
Change in child and parent relationship | From enrollment to the end of treatment at 4-6 months
  1 indicates the lowest scores and 5 indicates the highest scores in closeness and conflicts

SECONDARY OUTCOMES:
Change in synergy impact of inter-sectors | From enrollment to the end of treatment at 4-6 months
  1 indicates the lowest score and 5 indicates the highest scores in synergy impact

CONTACTS AND LOCATIONS:
Overall Officials: Anna Hui, PhD, Principal Investigator — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
It is because the participants do not give right to share their data with researchers not in the study.

REFERENCES:
- [Background] Leung C, Hui ANN, Wong RS, Rao N, Karnilowicz W, Chung K, Chan J, Ip P. Effectiveness of a Multicomponent Parenting Intervention for Promoting Social-Emotional School Readiness Among Children From Low-Income Families in Hong Kong: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2022 Apr 1;176(4):357-364. doi: 10.1001/jamapediatrics.2021.6308. PMID 35129606
- See also: This is the homepage of the project operated by the funder. — https://www.keysteps.hk/en/home